CLINICAL TRIAL: NCT02963428
Title: Teaching Appropriate Gestational Weight Gain
Acronym: TAGG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Penn State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-0205
Record Dates: First submitted 2016-10-12; First posted 2016-11-15 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Participants will receive the usual standard of care which includes written educational materials as well as counseling by their obstetric care provider.
- Enhanced Care (EC) (Experimental): In addition to standard of care, the study participants will also receive:
  i. An initial consult with a licensed, Registered Dietician Nutritionist (RDN); ii. Regular tele-health check-ups (10-20 mins/check-up) with the RDN until delivery; iii. Exposure to personal GWG chart; iv. Letter from physician stating the recommendations for GWG over the course of the pregnancy.
  Interventions: Behavioral: Enhanced Care

INTERVENTIONS:
Behavioral: Enhanced Care — In addition to standard of care, the study participants will also receive:
  i. An initial consult with a licensed, Registered Dietician Nutritionist (RDN); ii. Regular tele-health check-ups (10-20 mins/check-up) with the RDN until delivery; iii. Exposure to personal GWG chart; iv. Letter from physician stating the recommendations for GWG over the course of the pregnancy.
  Other Names: EC
  Arms: Enhanced Care (EC)

SUMMARY:
The study aims to improve obstetrical care by managing gestational weight gain (GWG) among high risk women in an effort to reduce maternal and fetal complications.

DETAILED DESCRIPTION:
The project is aimed at teaching women about the appropriate weight gain during pregnancy to optimize health outcomes for mothers and newborn babies. Obese gravida meeting inclusion criteria and none of the exclusion criteria will be offered enrollment in TAGG. Those that consent will be randomized to receive standard of care or enhanced care regarding gestational weight gain.

The primary outcome is the proportion of patients that gain less than 20 lbs over the course of the pregnancy. Secondary outcomes include patient knowledge and expectations, attitude about pregnancy weight gain, self-efficacy of ability to eat healthy, and eating, sleeping and physical activity behavior, perceived stress, psychological factors, patient-experience, involvement in care, and food security.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pregnancy body mass index of at least 30 kg/m2 (per patient report of weight)
* Less than 16 weeks gestation
* Gestational weight gain (GWG) less than < 11 pounds from their pre-pregnancy weight to time of potential study enrollment
* Singleton gestation
* Access to a phone

Exclusion Criteria:

* BMI less than 30 kg/m2
* Gestational age greater than or equal to 16 weeks
* Active diagnosis of cancer on their electronic health record problem list
* Acquired immunodeficiency syndrome (AIDS)
* Palliative medicine patients
* Multiple gestations
* GWG in excess of 11 pounds prior to study enrollment
* Patients with Non-Geisinger prenatal care providers
* Vegan diet
* Malabsorptive conditions
* Previously enrolled in TAGG during prior pregnancy. Patient will be excluded from re-randomization
* Non-English Speaking

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-11; Primary Completion 2018-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain, adjusting for time in the study | at delivery

SECONDARY OUTCOMES:
Patient knowledge and expectations factors | Baseline, 32-34 Weeks Gestation, and 4-12 Weeks Postpartum
  Participants will be enrolled at baseline (Less than 16 6/7 weeks gestation) and be given a self-report survey tool developed using validated instruments to complete assessing these constructs. This survey tool will then be administered at 32-34 weeks gestation and 4-12 postpartum assessing end of pregnancy and post-intervention patient knowledge and expectations factors.
Attitude on pregnancy weight gain | Baseline, 32-34 Weeks Gestation, and 4-12 Weeks Postpartum
  Participants will be enrolled at baseline (Less than 16 6/7 weeks gestation) and be given a self-report survey tool developed using validated instruments to complete assessing these constructs. This survey tool will then be administered at 32-34 weeks gestation and 4-12 postpartum assessing end of pregnancy and post-intervention patient attitudes on pregnancy weight gain.
Self-efficacy of healthy eating | Baseline, 32-34 Weeks Gestation, and 4-12 Weeks Postpartum
  Participants will be enrolled at baseline (Less than 16 6/7 weeks gestation) and be given a self-report survey tool developed using validated instruments to complete assessing these constructs. This survey tool will then be administered at 32-34 weeks gestation and 4-12 postpartum assessing end of pregnancy and post-intervention patient self-efficacy of healthy eating.
Eating, sleeping and physical activity behavior | Baseline, 32-34 Weeks Gestation, and 4-12 Weeks Postpartum
  Participants will be enrolled at baseline (Less than 16 6/7 weeks gestation) and be given a self-report survey tool developed using validated instruments to complete assessing these constructs. This survey tool will then be administered at 32-34 weeks gestation and 4-12 postpartum assessing end of pregnancy and post-intervention patient eating, sleeping and physical activity behaviors.
Patient-experience and involvement in care | Baseline, 32-34 Weeks Gestation, and 4-12 Weeks Postpartum
  Participants will be enrolled at baseline (Less than 16 6/7 weeks gestation) and be given a self-report survey tool developed using validated instruments to complete assessing these constructs. This survey tool will then be administered at 32-34 weeks gestation and 4-12 postpartum assessing end of pregnancy and post-intervention patient experience and involvement in their care.
Delivery of large for gestational age infants | At Delivery
  This measure will be obtained using electronic health record data and analyzed utilizing clinic data points as well as information gathered from patients through self-report survey data.
Diagnosis of gestational diabetes mellitus | Baseline through 4-12 Weeks Postpartum
  This measure will be obtained using EHR data and analyzed utilizing clinic data points.
Neonatal intensive care unit (NICU) admissions | At Delivery
Cost of Treatment | Baseline through 4-12 Weeks Postpartum
  Participant cost of treatment will be assessed utilizing claims data obtained from Geisinger Health Plan to compare the effectiveness of the intervention in reducing cost.
Mode of delivery | At Delivery
  Clinical electronic health record data in regards to the participant mode of delivery will be utilized in statistical analyses to determine whether mode of delivery has an impact on other outcomes of interest.
Rate of gestational weight gain | Baseline through 4-12 weeks postpartum
Perceived stress measured via Perceived Stress Scale | Baseline through 4-12 weeks postpartum
  Perceived Stress will be measured using the Perceived Stress Scale by Cohen et. al.
Psychological factors measured via Pregnancy Weight Gain Attitude Scale | Baseline through 4-12 Weeks postpartum
  Psychological factors will be assessed using the Pregnancy Weight Gain Attitude Scale by Palmer et. al.

CONTACTS AND LOCATIONS:
Overall Officials: Awathif D Mackeen, MD, MPH, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided